CLINICAL TRIAL: NCT00016146
Title: Vaccination Of Prostate Cancer Patients With A Bivalent Vaccine Containing MUC-2 Glycopeptide And Globo H Conjugates: A Dose-Escalating Trial Studying The Immunogenicity And Safety Of The Immunological Adjuvant GPI-0100
Brief Title: Vaccine Therapy Plus Biological Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99-062; P30CA008748 (NIH); MSKCC-99062; NCI-G01-1941
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — GPI0100

ARMS (1):
- vaccine (Experimental): This is a dose-escalation study of GPI-0100.
  Patients receive glycosylated MUC-2-Globo H-KLH conjugate vaccine with adjuvant GPI-0100 subcutaneously weekly on weeks 0-2, 6, 14, and 26 in the absence of unacceptable toxicity or disease progression.
  Cohorts of 5 patients receive escalating doses of GPI-0100 until the optimal dose, based on antibody response, is reached.
  Patients are followed every 3 months.
  Interventions: Biological: GPI-0100; Biological: MUC-2-Globo H-KLH conjugate vaccine

INTERVENTIONS:
Biological: GPI-0100
Biological: MUC-2-Globo H-KLH conjugate vaccine

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing. Combining vaccine therapy with biological therapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness in combining vaccine therapy and biological therapy in treating patients who have relapsed prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the optimal (in terms of antibody response) and safe dose range of glycosylated MUC-2-Globo H-KLH conjugate vaccine with adjuvant GPI-0100 in patients with biochemically relapsed prostate cancer.
* Assess post-immunization changes in prostate-specific antigen levels and other objective parameters of disease in these patients.

OUTLINE: This is a dose-escalation study of GPI-0100.

Patients receive glycosylated MUC-2-Globo H-KLH conjugate vaccine with adjuvant GPI-0100 subcutaneously weekly on weeks 0-2, 6, 14, and 26 in the absence of unacceptable toxicity or disease progression.

Cohorts of 5 patients receive escalating doses of GPI-0100 until the optimal dose, based on antibody response, is reached.

Patients are followed every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer
* Biochemically progressive disease after primary surgery or radiotherapy with or without neoadjuvant androgen ablation

  * Greater than 50% increase in PSA level above baseline value of 1.0 ng/mL post-prostatectomy or 2.0 ng/mL post-radiotherapy, based on 3 successive determinations taken at 2-week intervals
* Patients with prior intermittent hormonal therapy and non-castrate levels of testosterone are eligible
* Evaluable disease
* No radiographic evidence of metastasis
* No active CNS or epidural tumor
* No soft tissue and/or bone disease
* No androgen-independence with no evidence of radiographic disease
* May not be symptomatic or anticipated to develop symptoms within 6 months of study entry
* Concurrent registration to protocol MSKCC-90-040 required

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* At least 6 months

Hematopoietic:

* WBC at least 3,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than 2.0 mg/dL OR
* SGOT less than 3 times upper limit of normal

Renal:

* Creatinine no greater than 2.0 mg/dL OR
* Creatinine clearance at least 40 mL/min

Cardiovascular:

* No clinically significant cardiac disease (New York Heart Association class III or IV)

Pulmonary:

* No severe debilitating pulmonary disease

Other:

* No other prior malignancy within the past 5 years except nonmelanoma skin cancer
* No positive stool guaiac except hemorrhoids or history of documented radiation-induced proctitis
* No narcotic-dependent pain
* No infection requiring antibiotics
* No requirement for immunosuppressive therapy
* No allergy to seafood

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* See Disease Characteristics
* At least 2 weeks since change in hormonal therapy (except to maintain castrate levels of testosterone), including prednisone or dexamethasone
* At least 8 weeks since prior suramin and/or documented plasma concentration
* of suramin is less than 50 micrograms/mL (replacement hydrocortisone allowed)

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy to only measurable lesion

Surgery:

* See Disease Characteristics
* No concurrent surgery of only measurable lesion

Other:

* Recovered from prior therapy
* No other concurrent oncolytic agents
* No concurrent immunosuppressive therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2000-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
safety | 2 years

SECONDARY OUTCOMES:
immune function | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Susan Slovin, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States